CLINICAL TRIAL: NCT02419469
Title: Augmented Berlin-Frankfurt-Munster Therapy Plus Ofatumumab for Young Adults With Acute Lymphoblastic Leukemia or Lymphoblastic Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0396; NCI-2015-00967 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2015-04-14; First posted 2015-04-17 (Estimated); Results first posted 2018-06-11 (Actual); Last update posted 2018-06-11 (Actual); Status verified 2018-05

CONDITIONS: Leukemia; Precursor-B Acute Lymphoblastic Leukemia; Lymphoblastic Lymphoma; Lymphoma
Keywords: Leukemia; Precursor-B acute lymphoblastic leukemia; ALL; Lymphoblastic lymphoma; LL; Lymphoma; Cytarabine; Ara-C; Cytosar; DepoCyt; Cytosine Arabinosine Hydrochloride; Daunorubicin; Daunorubicin Hydrochloride; Cerubidine; Daunomycin; DNR; Vincristine; Prednisone; PEG asparaginase; Pegaspargase; Oncaspar; Polyethylene glycol conjugated lasparaginase-H; Ofatumumab; Arzerra; Rituximab; Rituxan; Methotrexate; Cyclophosphamide; Cytoxan; Neosar; Mercaptopurine; 6-mercaptopurine; Purinethol; 6-MP; Doxorubicin; Doxorubicin hydrochloride; Adriamycin PFS; Adriamycin RDF; Adriamycin; Rubex; Dexamethasone; Decadron; Thioguanine; 6-thioguanine
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma | interventions — Cytarabine; Daunorubicin; Vincristine; Prednisone; pegaspargase; ofatumumab; Rituximab; Methotrexate; Cyclophosphamide; Mercaptopurine; Doxorubicin; dexamethasone acetate; Calcium Dobesilate; Thioguanine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Augmented BFM Therapy + Ofatumumab or Rituximab (Experimental): Participants receive the study drugs in Induction, Consolidation, and Maintenance Courses.
  Interventions: Drug: Cytarabine; Drug: Daunorubicin; Drug: Vincristine; Drug: Prednisone; Drug: PEG asparaginase; Drug: Ofatumumab; Drug: Rituximab; Drug: Methotrexate; Drug: Cyclophosphamide; Drug: Mercaptopurine; Drug: Doxorubicin; Drug: Dexamethasone acetate; Drug: Thioguanine

INTERVENTIONS:
Drug: Cytarabine — Participants initially receive intrathecal treatment using Cytarabine 100 mg on Day 1. Induction chemotherapy must begin within 3 days of the intrathecal Cytarabine dose.
  Consolidation Therapy 1: Cytarabine 75 mg/m2 subcutaneously Days 1 - 4 and 8 - 11.
  Consolidation Therapy 3B: Cytarabine 75 mg/m2 subcutaneously Days 1 - 4 and Days 8 - 11.
  Other Names: Ara-C; Cytosar; DepoCyt; Cytosine Arabinosine Hydrochloride
Drug: Daunorubicin — Induction Therapy: Daunorubicin 25 mg/m2 by vein weekly for 4 doses.
  Other Names: Daunorubicin Hydrochloride; Cerubidine; Daunomycin; DNR
Drug: Vincristine — Induction Therapy: Vincristine 1.5 mg/m2 by vein weekly for 4 doses.
  Consolidation Therapy 1: Vincristine 1.5 mg/m2 by vein Week 3 and Week 4.
  Consolidation Therapy 2: Vincristine 1.5 mg/m2 by vein every 10 days for 5 doses.
  Consolidation Therapy 3A: Vincristine 1.5 mg/m2 by vein weekly for 3 doses.
  Consolidation Therapy 3B: Vincristine 1.5 mg/m2 by vein Weeks 3 and 4.
  Maintenance Therapy (24 months): Vincristine 1.5 mg/m2 by vein every 28 days.
Drug: Prednisone — Induction Therapy: Prednisone 60 mg/m2/day by mouth for 28 days.
Drug: PEG asparaginase — Induction Therapy: PEG asparaginase 2000 IU/m2 by vein on Day 4 of induction.
  Consolidation Therapy 1: PEG-asparaginase 2000 IU/m2 by vein Week 3 and Week 7.
  Consolidation Therapy 2: PEG-asparaginase 2000 IU/m2 by vein Weeks 1 and 4.
  Consolidation Therapy 3A: PEG-asparaginase 2000 IU/m2 by vein in Week 1.
  Consolidation Therapy 3B: PEG-asparaginase 2000 IU/m2 by vein Week 3.
  Other Names: Pegaspargase; Oncaspar; Polyethylene Glycol Conjugated Lasparaginase-H
Drug: Ofatumumab — Induction Therapy: Ofatumumab 300 mg by injection or vein on Day 2 and Ofatumumab 2000 mg by injection or vein on Day 15.
  Consolidation Therapy 1: Ofatumumab 2000 mg by injection or vein Week 1 and Week 5.
  Consolidation Therapy 2: Ofatumumab 2000 mg by injection or vein Week 1 and Week 5.
  Consolidation Therapy 3A: Ofatumumab 2000 mg by injection or vein Week 1 and Week 3.
  Other Names: Arzerra
Drug: Rituximab — Induction Therapy: If Ofatumumab not available, Rituximab 375 mg/m2 by vein on Day 1 and on Day 15.
  Consolidation Therapy 1: If Ofatumumab not available, Rituximab 375 mg/m2 by vein Week 1 and Week 5.
  Consolidation Therapy 2: If Ofatumumab not available, Rituximab 375 mg/m2 by vein Week 1 and Week 5.
  Consolidation Therapy 3A: If Ofatumumab not available, Rituximab 375 mg/m2 by vein Week 1 and Week 3.
  Other Names: Rituxan
Drug: Methotrexate — Induction Therapy: Intrathecal methotrexate 12 mg on Day 8 and Day 29.
  Consolidation Therapy 1: Intrathecal methotrexate 12 mg Weekly, Weeks 1 - 4.
  Consolidation Therapy 2: Methotrexate by vein every 10 days starting at 100 mg/m2 and increasing by 50 mg/m2 as tolerated. and Intrathecal methotrexate 12 mg Week 1.
  Consolidation Therapy 3A: Intrathecal methotrexate 12 mg in Week 1.
  Consolidation Therapy 3B: Intrathecal methotrexate 12 mg Week 1 and 2.
  Maintenance Therapy (24 months): Methotrexate 20 mg/m2 by mouth weekly, hold on days of intrathecal methotrexate.
  Maintenance Therapy (24 months): Intrathecal methotrexate 12 mg every 3 months for 4 doses.
Drug: Cyclophosphamide — Consolidation Therapy 1: Cyclophosphamide 1 gram/m2 by vein Week 1 and Week 5.
  Consolidation Therapy 3B: Cyclophosphamide 1 gram/m2 by vein Week 1.
  Other Names: Cytoxan; Neosar
Drug: Mercaptopurine — Consolidation Therapy 1: Mercaptopurine 60 mg/m2/day by mouth Days 1 - 14.
  Maintenance Therapy (24 months): Mercaptopurine 75 mg/m2 by mouth nightly.
  Other Names: 6-Mercaptopurine; Purinethol; 6-MP
Drug: Doxorubicin — Consolidation Therapy 3A: Doxorubicin 25 mg/m2 by vein weekly for 3 doses.
  Other Names: Doxorubicin Hydrochloride; Adriamycin PFS; Adriamycin RDF; Adriamycin; Rubex
Drug: Dexamethasone acetate — Consolidation Therapy 3A: Dexamethasone 10 mg/m2 by mouth on Days 1 - 7 and Days 15 - 21.
  Maintenance Therapy (24 months): Dexamethasone 6 mg/m2/day by mouth Days 1 - 5 every 28 days.
  Other Names: Decadron
Drug: Thioguanine — Consolidation Therapy 3B: Thioguanine 60 mg/m2/day by mouth for 14 days.
  Other Names: 6-thioguanine

SUMMARY:
The goal of this clinical research study is to learn if a chemotherapy combination called augmented Berlin-Frankfurt-Munster (BFM), when also combined with ofatumumab or rituximab, can help to control precursor-B ALL or LL in patients who are 12-30 years of age. The safety of these drug combinations will also be studied.

Augmented BFM is made up of daunorubicin, vincristine, prednisone, dexamethasone, PEG asparaginase, and methotrexate.

DETAILED DESCRIPTION:
Study Drug Administration:

If you are found to be eligible to take part in this study, on Day 1 or during the spinal tap procedure, you will be given cytarabine as an injection in your spinal fluid.

You will then receive the study drugs in Induction, Consolidation, and Maintenance Courses. Induction Therapy is designed to remove the signs of leukemia that can be seen and to allow normal blood cells to be restored. This is called remission. Consolidation and Maintenance Therapies are designed to cause the disease to stay in remission.

The study drugs will be given the following ways:

* Daunorubicin by vein over about 30 minutes
* Vincristine by vein over 15-30 minutes
* PEG asparaginase by vein over 15-60 minutes
* Methotrexate either by mouth or as an injection into your spinal fluid (intrathecal), depending on the course. When given through the spinal fluid, cerebrospinal fluid (CSF) will be collected with each spinal tap to test the fluid for leukemia. If there is disease in your spinal fluid before starting the treatment, you will be given additional methotrexate doses each week until there is no disease present.
* Ofatumumab as an injection or by vein. If given by vein, the length of the infusion will depend on how well you tolerate the drug. If ofatumumab is not available, you will be given rituximab by vein over several (about 4-6) hours.
* Cyclophosphamide by vein over about 1 hour
* Cytarabine as an injection under the skin or by vein. If given by vein, the length of the infusion will depend on how well you tolerate the drug.
* Doxorubicin by vein. If given by vein, the length of the infusion will depend on how well you tolerate the drug.
* Prednisone, 6-Mercaptopurine, dexamethasone, and 6-Thioguanine are all taken by mouth

Within 3 days after you receive cytarabine, you will begin the Induction Course, which will last for 4 weeks. In the Induction Course, you will receive:

* Daunorubicin and vincristine on Days 1, 8, 15, and 22
* PEG asparaginase 1 time during Week 1
* Prednisone each day on Days 1-28.
* Intrathecal methotrexate at Weeks 2 and 5 during a spinal tap. If the is disease in your spinal fluid before starting the treatment, you will be given additional methotrexate doses each week until there is no disease present.
* Ofatumumab or rituximab on Days 2 and 15

Depending on how you respond to Induction, you may begin the Consolidation Courses 1-4 weeks after Induction.

You will then receive Consolidation Course 1. This course will last 8 weeks, and you will receive:

* Cyclophosphamide at Weeks 1 and 5
* Cytarabine on or around Days 1-4 and Days 8-11 of each 4-week cycle
* 6-Mercaptopurine on Days 1-14 of each 4-week cycle
* Vincristine at Weeks 3 and 4 of each 4-week cycle
* PEG Asparaginase at Weeks 3 and 7
* Intrathecal methotrexate weekly during Month 1 only
* Ofatumumab or rituximab at Weeks 1 and 5

You will then receive 2 courses of Consolidation Course 2. Each course will last about 7 weeks, and you will receive:

* Vincristine and methotrexate every 10 (+/- 2) days for up to 5 doses
* PEG Asparaginase at Weeks 1 and 4
* Intrathecal methotrexate at Weeks 1 and 5
* Ofatumumab or rituximab at Weeks 1 and 5

You will then receive Consolidation 3 (Part A). This course will last for 4 weeks, and you will receive:

* Vincristine and doxorubicin at Weeks 1, 2, and 3
* Dexamethasone on Days 1-7 and Days 15-21
* PEG asparaginase at Week 1
* Intrathecal methotrexate at Week 1
* Ofatumumab or rituximab on Weeks 1 and 3

You will then receive Consolidation 3 (Part B). This course will last for 4 weeks, and you will receive:

* Cyclophosphamide at Week 1
* Cytarabine for 4 days in a row during Weeks 1-2
* 6-Thioguanine every day for the first 2 weeks.
* Intrathecal methotrexate at Weeks 1 and 2
* Vincristin at Weeks 3 and 4
* PEG Asparaginase at Week 3

Once you finish Consolidation, you will then receive 24 months of Maintenance Therapy.

* Vincristine every month.
* Dexamethasone for 5 days every month.
* 6-Mercaptopurine 1 time a day
* Methotrexate by mouth every week.
* If you have ALL, you will also receive intrathecal methotrexate every 3 months for the first 12 months of maintenance.

Study Tests/Procedures:

Induction:

* Blood (about 3 teaspoons) will be drawn about 2 times each week during the Induction Period for routine tests.
* You will have a bone marrow aspirate or biopsy on Days 15 and 29 and then as needed to check the status of the disease.
* About 7 days after you receive your first dose of PEG asparaginase, blood (about 1 tablespoon) will be drawn to check the activity of the drug in your blood. If the drug does not seem to be working well, your dose may be changed.
* If you have LL and bone marrow was not found to be involved with the disease at screening, you will have a chest x-ray, CT scans, and positron emission tomography (PET) scans to measure the disease. These scans will be done after about 28 days of therapy.

Consolidation 1:

* Blood (about 3 teaspoons) will be drawn for routine tests about 2 times each week.
* You will have a spinal tap during each intrathecal methotrexate dose. The spinal fluid will be checked for leukemia cells.
* You will have a bone marrow aspiration at the end of Month 2 to check the status of the disease.

Consolidation 2:

* Blood (about 3 teaspoons) will be drawn every 2 weeks for routine tests.
* You will have a spinal tap during each intrathecal methotrexate doses. The spinal fluid will be checked for leukemia cells.

Consolidation 3 (Part A and B):

* Blood (about 3 teaspoons) will be drawn at least weekly for routine tests.
* You will have a spinal tap during each intrathecal methotrexate dose. The spinal fluid will be checked for leukemia cells.

Maintenance:

* You will have a spinal tap during each intrathecal methotrexate dose. The spinal fluid will be checked for leukemia cells.
* You will have a bone marrow aspiration at least every 3-6 months to check the status of the disease.

Length of Study:

You may remain on study for as long as the study doctor thinks it is in your best interest. If the disease does not appear to be improving after Induction, you will be taken off study. You may be taken off study if the disease gets worse or comes back during treatment, if intolerable side effects occur, if your doctor thinks it is in your best interest, or if you cannot follow the study instructions.

Follow-up Visits:

Your study doctor will inform you of your follow-up visit schedule in the clinic. At each follow-up visit there will be a physical exam and blood (about 1 tablespoon) will be drawn for routine tests. You will be followed-up for the next 3 years after your the last dose of your chemotherapy.

This is an investigational study. The chemotherapy drugs used in this study are all FDA approved and commercially available for the treatment of various types of leukemia. The use of ofatumumab/rituximab in this drug combination, as well as the drug combination's use in pediatric patients, is investigational.

Up to 100 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have precursor-B lymphoblastic leukemia or lymphoma.
2. Patients must be untreated or have had only one prior chemotherapy regimen for ALL or LL . Previously treated patients will be analyzed separately.
3. Age between 12 to 30 years old
4. Patients with central nervous system (CNS) disease or testicular disease are eligible.
5. Intrathecal therapy with cytarabine is allowed prior to registration for patient convenience. This is usually done at the time of the diagnostic bone marrow or venous line placement to avoid a second lumbar puncture. Systemic chemotherapy must begin within 72 hours of the first intrathecal treatment.
6. Signed informed consent prior to the start of systemic therapy. In the event of enrollment of a minor patient, an attempt to obtain assent from the patient must be documented, and parental consent must be signed.
7. Echocardiogram should be done within 7 days of starting therapy if there are cardiac risk factors (e.g., history of hypertension or of myocardial infarction)
8. Creatinine should be < 3 mg/dL bilirubin < 3 mg/dl unless due to disease
9. Zubrod Performance status of <3
10. Patients who received steroids more than 72 hours prior to study enrollment are eligible but will be analyzed separately.
11. Lymphoblasts may have any positive expression of cluster of differentiation antigen 20 (CD20) for ofatumumab administration.

Exclusion Criteria:

1. Age less than twelve years of age or greater than 30 years.
2. More than one prior treatment regimen for ALL or LL.
3. The patient is pregnant or unwilling to practice appropriate birth control.
4. Presence of the Philadelphia chromosome t(9;22)
5. Laboratory or clinical evidence of active infectious hepatitis.

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2015-11-13 (Actual); Primary Completion 2017-06-22 (Actual); Study Completion 2017-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael E. Rytting, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Ofatumumab Plus Chemotherapy: Ofatumumab plus chemotherapy. Only one patient enrolled prior to termination.
Period: Overall Study
Arm/Group | Ofatumumab Plus Chemotherapy
Started | 1
Completed | 0
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ofatumumab Plus Chemotherapy
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Event Free Survival (EFS)
Description: Event free survival defined as the time from treatment to relapse of leukemia or death for any reason or lost to follow-up. Study regimen considered successful if it exhibits a 3-year EFS rate greater than 65% and response rate no less than 90% with Grade III-IV infectious toxicity rate in induction no more than 33%.
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Ofatumumab Plus Chemotherapy
Number analyzed (Participants) | 1
Participants | NA — Participant was lost to follow up.

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Ofatumumab Plus Chemotherapy
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-12): https://cdn.clinicaltrials.gov/large-docs/69/NCT02419469/Prot_SAP_000.pdf